CLINICAL TRIAL: NCT00164931
Title: Phase 3 Study of Prospective Randomized Trial Comparing Adjunctive High Dose Omeprazole Infusion Against Scheduled Second Endoscopy in the Prevention of Peptic Ulcer Rebleeding After Therapeutic Endoscopy
Brief Title: A Study Comparing High Dose Omeprazole Infusion Against Scheduled Second Endoscopy for Bleeding Peptic Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCHCE03-43-SURG5
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2005-09

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic ulcer hemorrhage; Omeprazole; Scheduled second endoscopy
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

INTERVENTIONS:
Drug: Intravenous omeprazole infusion
Procedure: Scheduled second endoscopy

SUMMARY:
A prospective randomized study to compare the adjunctive use of high dose omeprazole infusion against scheduled second endoscopy in prevention of peptic ulcer rebleeding after therapeutic endoscopy.

DETAILED DESCRIPTION:
We have previously performed a prospective randomized controlled trial on the effect of scheduled second endoscopy upon peptic ulcer rebleeding. We found that the rate of recurrent bleeding was significantly reduced from 13.8% to 5% with a scheduled second endoscopy and appropriate therapy performed within 24 hours after initial hemostasis.

When we look at the studies in the literature employing proton pump inhibitors (PPI) infusion after primary endoscopic therapy, we found that there was also a significant reduction in the rate of rebleeding, the number of operation performed and the transfusion requirement.

Controversy exists regarding the optimal strategy to minimize recurrent peptic ulcer bleeding after successful endoscopic hemostasis. A recent cost-effective analysis on various strategies showed that selective scheduled second endoscopy strategy was probably the most effective and least expensive to prevent recurrent peptic ulcer bleeding.

We conduct a randomized trial on the cost-effectiveness of using omeprazole infusion vs scheduled second endoscopy on the management of bleeding peptic ulcers.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients admitted for peptic ulcer bleeding (including bleeding anastomotic ulcers) with emergency endoscopy done in 24 hours after admission with Forrest type Ia, Ib, and IIa, IIb
* age 15 - 90 years
* Written consent available

Exclusion Criteria:

* ulcer bleeding not controlled in first endoscopy
* Bleeding from malignant ulcer or tumor
* Bleeding from Dieulafoy lesion/ angiodysplasia
* Bleeding from injection sclerotherapy ulcer
* Patient with ASA category 5

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2003-10

PRIMARY OUTCOMES:
Recurrent bleeding within 30 days after initial endoscopy defined as -
Clinical criteria (anyone of the below)
1. Haemetmesis or fresh blood from Ryles tube
2. Fresh melena with shock (systolic blood pressure < 100mmHg or pulse >100/min) or drop in Hb > 2g/dl
3. Haemoglobin drop for more than 4 g/dl in 24 hours before 2nd therapeutic endoscopy
4. Blood transfusion of > 4 unit in 24 hours to stabilize Hb level or vital signs
AND Endoscopic criteria of Forrest I a, b or II a, b

SECONDARY OUTCOMES:
1. The rate of surgery
2. Mortality
3. Length of Hospital stay
4. Transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Philip WY Chiu, MBChB, FRCSEd, Principal Investigator — Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong; Henry KM Joeng, MBBS, Principal Investigator — Department of Surgery, United Christian Hospital, Hong Kong
Locations (1):
- Department of Surgery, United Christian Hospital, Hong Kong, China